CLINICAL TRIAL: NCT04241653
Title: Impact of Different Modes of Ventilation With Laryngeal Mask Airway on Pediatric Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sameh Fathy (Other)
Responsible Party: Sponsor-Investigator, Sameh Fathy, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ventilation with LMA
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Ventilation; Laryngeal Mask Airway; Cataract Surgery
MeSH Terms: conditions — Respiratory Aspiration | interventions — Ventilation; Positive-Pressure Respiration; Laryngeal Masks; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spontaneous Ventilation (Active Comparator): Patients will spontaneously ventilated. Laryngeal mask airway will be inserted and anesthesia is maintained with sevoflurane.
  Interventions: Procedure: Pressure Support Ventilation; Device: Laryngeal Mask Airway; Drug: Sevoflurane
- Unparalyzed Controlled Ventilation (Active Comparator): Patients will be mechanically ventilated without muscle relaxation.Laryngeal mask airway will be inserted and anesthesia is maintained with sevoflurane.
  Interventions: Procedure: Unparalyzed Pressure Control Ventilation; Device: Laryngeal Mask Airway; Drug: Sevoflurane
- Paralyzed Controlled Ventilation (Active Comparator): Patients will be mechanically ventilated with muscle relaxation.Laryngeal mask airway will be inserted and anesthesia is maintained with sevoflurane.
  Interventions: Procedure: Paralyzed Pressure Control Ventilation; Device: Laryngeal Mask Airway; Drug: Sevoflurane

INTERVENTIONS:
Procedure: Pressure Support Ventilation — Ventilator will be adjusted to administer pressure at 10 cmH2O.
  Other Names: Assisted Ventilation
  Arms: Spontaneous Ventilation
Procedure: Unparalyzed Pressure Control Ventilation — Pressure controlled ventilation mode will be applied to obtain a volume of 8 ml/kg up to 20 cmH2O. The set respiratory rate will be 15 breaths/min then it is adjusted to achieve the end tidal CO2 levels between 35 and 40 mmHg as measured by capnography.
  Other Names: Positive pressure Ventilation
  Arms: Unparalyzed Controlled Ventilation
Procedure: Paralyzed Pressure Control Ventilation — Pressure controlled ventilation mode will be applied to obtain a volume of 8 ml/kg up to 20 cmH2O. The set respiratory rate will be 15 breaths/min then it is adjusted to achieve the end tidal CO2 levels between 35 and 40 mmHg as measured by capnography. Also, neuromuscular blockade will be achieved.
  Other Names: Positive pressure Ventilation
  Arms: Paralyzed Controlled Ventilation
Device: Laryngeal Mask Airway — Capnography connected to laryngeal mask airway is introduced after adequate jaw relaxation; its size is chosen according to the body weight of the child.
  Other Names: Supraglottic Airway Device
Drug: Sevoflurane — Sevoflurane in air/oxygen mixture of 40% will be titrated to achieve adequate depth of anesthesia to maintain immobilization of the eye.
  Other Names: Inhalational Anesthesia

SUMMARY:
This study will be conducted to evaluate effects of different modes of ventilation on pediatric cataract surgery aiming to a peri-operative stable anesthesia, better surgical satisfaction and post operative recovery. It is hypothesized that controlled ventilation without muscle relaxation will be advantageous to other modes in providing adequate surgical satisfaction with considerable depth of anesthesia and better recovery profile.

DETAILED DESCRIPTION:
Anesthetic management in pediatric cataract surgery constitutes a special challenge. Any eye movements can lead to an unsatisfactory surgical field and increase the risk of ophthalmological complications. Achieving adequate ventilation of children is considered another challenge due to huge variability in size and lung maturity. Spontaneous breathing is a popular mode of ventilation with several beneficial effects. Controlled ventilation without muscle relaxation using laryngeal mask airway is attractive option because the side effects of muscle relaxants are avoided. Therefore, this study will be conducted to evaluate effects of different modes of ventilation on pediatric cataract surgery aiming to a peri-operative stable anesthesia, better surgical satisfaction and post-operative recovery. This prospective, randomized, comparative clinical study will include 150 children who will be scheduled for elective cataract surgery under general anesthesia in Mansoura ophthalmology center over one year. Informed written consent will be obtained from parents of all subjects in the study after ensuring confidentiality.The study protocol will be explained to parents of all patients in the study who will be kept fasting prior to surgery. Patients will be randomly assigned to three equal groups according to computer-generated table of random numbers using the permuted block randomization method. In the first group, spontaneous ventilation will be maintained with pressure support; while in the two other groups, mechanical ventilation will be applied with pressure controlled modes. The collected data will be coded, processed, and analyzed using SPSS program. All data will be considered statistically significant if P value is ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I and II patients.
* Scheduled for elective cataract surgery.

Exclusion Criteria:

* Parental refusal of consent.
* Contraindication to use of supraglottic airway device as gastroesophageal reflux and oropharyngeal pathology.
* Hyperactive airway disease or respiratory diseases.
* Children with developmental delays, mental or neurological disorders.
* Bleeding or coagulation diathesis.
* History of known sensitivity to the used anesthetics.
* Previous surgery in the same eye.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Incidence of eye movements | Up to the end of the surgery
  Incidence any upward or downward deviation of the vision axis during surgery will be recorded

SECONDARY OUTCOMES:
Changes in intraocular pressure | Up to the end of the surgery
  Intraocular pressure will be measured (mmHg) in the non-operative eye using Schioetz-Tonometer
Changes in bispectral index | Up to the end of the surgery
  Bispectral index values (0-100) will be recorded every five minutes until the end of the surgery
Amount of consumption of sevoflurane | Up to the end of the surgery
  Sevoflurane consumption in milliliters will be measured and recorded
Changes in dynamic compliance | Up to the end of the surgery
  Dynamic compliance (ml /cm H2O) will be recorded after stabilization of ventilation and at the end of surgery
Changes in heart rate | Up to the end of the surgery
  Heart rate (beat/min) will be recorded at five-minute intervals until the end of the surgery
Changes in mean arterial blood pressure | Up to the end of the surgery
  Blood pressure (mmHg) will be recorded at five-minute intervals until the end of the surgery
Value of surgeon satisfaction from the procedure | After the end of the surgery
  The ophthalmogist will be investigated postoperatively for the quality of surgical field (0-8; 0=None, 8=total satisfaction)
Improvement in postoperative emergence agitation scale | Up to 30 minutes after surgery
  Agitation will be assessed using the 5- step Cravero scale (1-5) every five minutes from awakening and for 30 minutes. (1:Obtunded with no response to stimulation, 2:Asleep but responsive to movement or stimulation, 3:Awake and responsive, 4:Crying, 5:Thrashing behaviour that requires restraint)

CONTACTS AND LOCATIONS:
Overall Officials: Sameh M El-Sherbiny, MD, Study Director — Mansoura Faculty of Medicine
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dias R, Dave N, Agrawal B, Baghele A. Correlation between bispectral index, end-tidal anaesthetic gas concentration and difference in inspired-end-tidal oxygen concentration as measures of anaesthetic depth in paediatric patients posted for short surgical procedures. Indian J Anaesth. 2019 Apr;63(4):277-283. doi: 10.4103/ija.IJA_653_18. PMID 31000891
- [Background] Fudickar A, Gruenewald M, Fudickar B, Hill M, Wallenfang M, Hullemann J, Voss D, Caliebe A, Roider JB, Steinfath M, Treumer F. Immobilization during anesthesia for vitrectomy using a laryngeal mask without neuromuscular blockade versus endotracheal intubation and neuromuscular blockade. Minerva Anestesiol. 2018 Jul;84(7):820-828. doi: 10.23736/S0375-9393.17.12282-0. Epub 2017 Oct 12. PMID 29027777
- [Background] Ghabach MB, El Hajj EM, El Dib RD, Rkaiby JM, Matta MS, Helou MR. Ventilation of Nonparalyzed Patients Under Anesthesia with Laryngeal Mask Airway, Comparison of Three Modes of Ventilation: Volume Controlled Ventilation, Pressure Controlled Ventilation, and Pressure Controlled Ventilation-volume Guarantee. Anesth Essays Res. 2017 Jan-Mar;11(1):197-200. doi: 10.4103/0259-1162.200238. PMID 28298784
- [Background] Lewis SR, Pritchard MW, Fawcett LJ, Punjasawadwong Y. Bispectral index for improving intraoperative awareness and early postoperative recovery in adults. Cochrane Database Syst Rev. 2019 Sep 26;9(9):CD003843. doi: 10.1002/14651858.CD003843.pub4. PMID 31557307
- [Background] Waldschmidt B, Gordon N. Anesthesia for pediatric ophthalmologic surgery. J AAPOS. 2019 Jun;23(3):127-131. doi: 10.1016/j.jaapos.2018.10.017. Epub 2019 Apr 14. PMID 30995517
- [Background] Singh PM, Trikha A, Sinha R, Borle A. Measurement of consumption of sevoflurane for short pediatric anesthetic procedures: Comparison between Dion's method and Dragger algorithm. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):516-20. doi: 10.4103/0970-9185.119160. PMID 24249990
- [Background] Mason KP. Paediatric emergence delirium: a comprehensive review and interpretation of the literature. Br J Anaesth. 2017 Mar 1;118(3):335-343. doi: 10.1093/bja/aew477. PMID 28203739